CLINICAL TRIAL: NCT02964351
Title: microRNA Profiles Identification in Adeno Carcinoma Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Natalia Goldberg, Principal Investigator, Assuta Medical Center
Other Study IDs: 0093-16-ASMC
Record Dates: First submitted 2016-11-08; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Carcinosarcoma
Keywords: MicroRNA; Prostate Carcinoma; PET-MR
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — MicroRNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High PSA (prostate-specific antigen) levels
  Interventions: Biological: High PSA levels

INTERVENTIONS:
Biological: High PSA levels

SUMMARY:
In our study, the investigators want to find correlation between circulating miRNAs associated with prostate cancer metastases to bones and to lymph nodes separately with results of 68Ga-PSMA ligand PET (positron emission computed) imaging.

ELIGIBILITY:
Inclusion Criteria:

* Proven Adeno-carcinoma
* Underwent prostatectomy and still present high PSA levels
* Refered to PSMA exam.

Exclusion Criteria:

* Below 18 years old
* HIV/HBV (hepatitis B virus)/HCV (hepatitis C virus) positive
* Additional malignancy during the past five years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high PSA levels
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Metastasis size and location | 18 months
  Location of metastasis by a report analyzing the pathological examination (PET-MR output).

SECONDARY OUTCOMES:
MicroRNA profile by using Nano-string technology validated by real time PCR | 24 months
  Validation of MicroRNA pattern by using real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Goldberg, MD, Principal Investigator — Assuta Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berindan-Neagoe I, Monroig Pdel C, Pasculli B, Calin GA. MicroRNAome genome: a treasure for cancer diagnosis and therapy. CA Cancer J Clin. 2014 Sep-Oct;64(5):311-36. doi: 10.3322/caac.21244. Epub 2014 Aug 7. PMID 25104502
- [Background] Hovels AM, Heesakkers RA, Adang EM, Jager GJ, Strum S, Hoogeveen YL, Severens JL, Barentsz JO. The diagnostic accuracy of CT and MRI in the staging of pelvic lymph nodes in patients with prostate cancer: a meta-analysis. Clin Radiol. 2008 Apr;63(4):387-95. doi: 10.1016/j.crad.2007.05.022. Epub 2008 Feb 4. PMID 18325358
- [Background] Briganti A, Abdollah F, Nini A, Suardi N, Gallina A, Capitanio U, Bianchi M, Tutolo M, Passoni NM, Salonia A, Colombo R, Freschi M, Rigatti P, Montorsi F. Performance characteristics of computed tomography in detecting lymph node metastases in contemporary patients with prostate cancer treated with extended pelvic lymph node dissection. Eur Urol. 2012 Jun;61(6):1132-8. doi: 10.1016/j.eururo.2011.11.008. Epub 2011 Nov 12. PMID 22099610
- [Background] Weilbaecher KN, Guise TA, McCauley LK. Cancer to bone: a fatal attraction. Nat Rev Cancer. 2011 Jun;11(6):411-25. doi: 10.1038/nrc3055. Epub 2011 May 19. PMID 21593787
- [Background] Logothetis CJ, Lin SH. Osteoblasts in prostate cancer metastasis to bone. Nat Rev Cancer. 2005 Jan;5(1):21-8. doi: 10.1038/nrc1528. PMID 15630412
- [Background] Afshar-Oromieh A, Zechmann CM, Malcher A, Eder M, Eisenhut M, Linhart HG, Holland-Letz T, Hadaschik BA, Giesel FL, Debus J, Haberkorn U. Comparison of PET imaging with a (68)Ga-labelled PSMA ligand and (18)F-choline-based PET/CT for the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2014 Jan;41(1):11-20. doi: 10.1007/s00259-013-2525-5. Epub 2013 Sep 27. PMID 24072344
- [Background] Schmid DT, John H, Zweifel R, Cservenyak T, Westera G, Goerres GW, von Schulthess GK, Hany TF. Fluorocholine PET/CT in patients with prostate cancer: initial experience. Radiology. 2005 May;235(2):623-8. doi: 10.1148/radiol.2352040494. PMID 15858102